CLINICAL TRIAL: NCT02767115
Title: Grape Seeds Extract Gel as an Adjunct to Scaling and Root Planing for the Treatment of Chronic Periodontitis: A Pilot Clinical Study
Brief Title: Grape Seeds Extract Gel as an Adjunct for the Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Mohammad Ramadan Rayyan, Assistant professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUGRP/2014/182
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSE mucoadhesive gel (Experimental): 2%GSE mucoadhesive gel administered in the periodontal pockets of GSE group at T0 and 3, 6, and 9 days after T0
  Interventions: Dietary Supplement: 2% GSE mucoadhesive gel
- Control mucoadhesive gel (Placebo Comparator): GSE free mucoadhesive gel administered in the periodontal pockets of Control group at T0 and 3, 6, and 9 days after T0
  Interventions: Other: GSE free mucoadhesive gel

INTERVENTIONS:
Dietary Supplement: 2% GSE mucoadhesive gel — 2% GSE mucoadhesive gel administered in periodontal pockets of GSE group at T0 and 3, 6, and 9 days after T0
  Arms: GSE mucoadhesive gel
Other: GSE free mucoadhesive gel — GSE free mucoadhesive gel administered in periodontal pockets of Control group at T0 and 3, 6, and 9 days after T0
  Arms: Control mucoadhesive gel

SUMMARY:
The aim of this study was to formulate a mucoadhesive gel of grapes seed extract (GSE) followed by short-term clinical study for the effectiveness of this gel onto the pocket depth (PD), plaque index (PI), gingival index (GI), and bleeding on probing (BOP) when applied in periodontal pockets as an adjunct treatment for chronic periodontitis.

DETAILED DESCRIPTION:
Before commencing with the study, the trial proposal was registered in the research center and ethical clearance was taken from the ethical committee (FUGRP/2014/182)

Materials used in the study::

1. Pure Grape Seed Extract (GSE) supplied by pure bulk supplements (Bulksupplements, USA). It contains natural ingredient of more than 180 mg of proanthocyanidins for every 200 mg of serving size of the powder. GSE has been considered safe by the National Center for Complimentary and Integrative Health if used orally for up to 8 weeks of clinical trials
2. Carbapol "CB 934" (Loba Chemie Pvt. Ltd., Mumbai)
3. Sodium- carboxy methly cellulose "Na-CMC" supplied (Loba Chemie Pvt. Ltd., Mumbai)
4. Sodium phosphate monobasic and sodium phosphate dibasic (Acros organic Ltd., Mumbai)
5. Parabens (Loba Chemie Pvt. Ltd., Mumbai)

Method of preparation:

GSE mucoadhesive gel preparation:

- Formula 1: 2% GSE mucoadhesive gel based on minimum inhibitory concentration (MIC) and minimum toxic concentration (MTC) and depending on the concentration of adhesive polymers that were added to the formula.

Weighed CB 934 was dissolved in 50 ml of phosphate buffer of pH 6.6 with a vigorous mixing until it dissolved completely. Then, GSE and preservatives were dissolved in about 25 ml of phosphate buffer of pH 6.6. After that, the GSE solution was slowly added into the solution of CB 934 with a continuous stirring that was achieved by magnetic stirring at a speed of 100 rpm until a homogenous mixture was obtained. The gelling agent (Na-CMC) was added slowly under a continuous magnetic stirring. Then, the volume was increased up to 100 ml with the addition of phosphate buffer. Finally, the prepared gel was kept for 24 hours at room temperature (25°C) for a complete polymer dissolution.

- Formula 2: controlled gel without GSE. A controlled mucoadhesive gel was used in the clinical study to be compared with GSE gel. This control gel contained all above mentioned substances except for the GSE.

Microbial limit test:

One gram of the gel was suspended in 2.9 ml of phosphate buffer at pH 7.2. Different sterile media (Bismuth Sulfite Medium, Mannitol salt agar medium, Muller Hinton agar medium, cetrimide agar medium and sabaroud agar medium) were inoculated with the gel, then, incubated for 24 hours. After that, the media were examined to ensure no growth of bacterial genera.

Subjects:

A random sample of 24 patients were screened and examined. Five patients with mean age 43.5 ±7.9 years were found to comply with the study inclusion criteria

Baseline measurements and application of gels A total of 86 Sites of pocket depth (PD) of 5 mm and above were identified. Sites were divided randomly by split mouth technique into two groups: Test group (GSE group) who will receive GSE mucoadhesive gel (N=48) and Control group who will receive the control gel (N=38). The two prepared formulas were placed in identical containers providing that neither the patient, nor the clinician were aware of which was applied on which quadrant of the mouth "i.e. double blinded study".

In the first visit, an informed written consent was obtained from all patients. scaling and root planing (SRP) were performed by the same calibrated examiner using an ultrasonic scaler (miniPiezon, EMS, Switzerland) and Gracey curettes (Hu-Friedy Mfg, USA). Seven days after, the patients were recalled for clinical examination and baseline measurement (T0) were taken for Plaque index (PI), Gingival index (GI), Pocket depth (PD), and bleeding on probing (BOP) by a single calibrated examiner. PD was measured using a manual probe (UNC 15). PI and GI were assessed according to Silness and Loe (1964). BOP was assessed within 30 seconds after probing. In the same visit, the examiner applied the two prepared formulas into two opposite quadrants using a disposable syringe with a 23-gauge needle. Patients were given oral hygiene instructions and were instructed not to drink or eat for a minimum of 3 hours, not to brush the area for 24 hours and not to use mouth wash during the course of treatment.

The patients were recalled again after 3, 6, and 9 days to reapply the two formulas in the examined sites by the same examiner.

Revaluation The first re-evaluation visit (T1) was after 28 days from the baseline measurements (T0). During this visit, the calibrated clinician measured and recorded PI, GI, PD, BOP for all examined sites.

The second re-evaluation visit (T2) was after 6 months from the baseline measurements (T0) and the same measurements were retaken for all sites.

Statistical Package for the Social Sciences (SPSS) v20 package (IBM Corp) was used for statistical analysis. Significance of the change in PI, GI, and PD within each group were determined using paired t-test while the significance of difference in the change between the two groups was determined using the independent t-test. The difference was considered statistically significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* being medically fit
* non-smokers
* has clinical diagnosis of chronic periodontitis with pockets depth of 5mm or greater along with evident radiographic bone Loss, and acceptance to provide an informed consent

Exclusion Criteria:

* pregnant patients
* breastfeeding mothers
* patients who are taking dietary supplements
* patients known to have grape's allergy
* patients with hypertension or bleeding disorders
* patients who have been under systemic or topical antibiotic treatments in the last 3 months
* smokers, and patients who are taking any medications that may interact with GSE

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pocket depth (PD) score | before application of the gel (baseline T0), 4 weeks after first application (T1), 6 months after first application (T2)
  PD will be measured for all sites and compared with PD scores at T0

SECONDARY OUTCOMES:
Change from baseline Plaque index (PI)score | before application of the gel (baseline T0), 4 weeks after first application (T1), 6 months after first application (T2)
  PI will be measured for all sites and compared with PI scores at T0
Change from baseline Gingival index (GI)score | before application of the gel (baseline T0), 4 weeks after first application (T1), 6 months after first application (T2)
  GI will be measured for all sites and compared with GI scores at T0
Change from baseline Bleeding on probing (BOP) | before application of the gel (baseline T0), 4 weeks after first application (T1), 6 months after first application (T2)
  BOP will be examined for all sites and number of sites with positive BOP will be compared with number of sites with positive BOP at T0

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Rayyan, MDS, Principal Investigator — Assistant professor; Tammam S Terkawi, MSc, Principal Investigator — Lecturer
Locations (1):
- Riyadh colleges of dentistry and pharmacy, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided